CLINICAL TRIAL: NCT06999213
Title: Lower Limb ExoNET: Development and Evaluation for Gait Assistance With Stroke Survivors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00223221
Record Dates: First submitted 2025-04-07; First posted 2025-05-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All participants will receive either intervention, but the order in which they receive it will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will receive Sham → Assist → Resist in a crossover design.
  Interventions: Other: Assist; Other: Resist; Other: Slack
- Group 2 (Experimental): Participants will receive Sham → Resist → Assist in a crossover design
  Interventions: Other: Assist; Other: Resist; Other: Slack

INTERVENTIONS:
Other: Assist — The device will provide assistive torques to support either ankle, knee, and/or hip movements.
Other: Resist — The device will apply resistive torques to exaggerate gait asymmetries, facilitating error augmentation.
  Other Names: Anti-Assistance
Other: Slack — The device will be worn but will not generate any torque.

SUMMARY:
Stroke-related gait impairments, such as poor limb coordination, imbalance, and reduced push-off strength, are often addressed using robotic systems or electrical stimulation, which can be costly, invasive, or insufficient for long-term recovery. Current devices often assist movement but fail to promote functional motor learning. Research supports rehabilitation strategies that amplify gait errors to drive neuroplasticity and adaptation. The LegExoNET (Exoskeletal Network for Elastic Torque) is a novel, passive wearable exoskeleton designed to address this need by enabling both assistive and therapeutic gait training. It stores and releases elastic energy to aid movement while allowing natural joint motion. The system aims to support individuals post-stroke transitioning to independent rehabilitation by offering a lightweight, affordable, and adaptive solution. Initial testing will focus on healthy individuals to assess safety and feasibility before expanding to stroke populations. The LegExoNET has the potential to enhance gait recovery and reduce therapist burden through error augmentation and personalized support, both in clinical and at-home settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Ability to provide informed consent
* Capable of ambulating without the use of assistive devices for 2 hours

Exclusion Criteria:

* History of stroke, SCI, or other neurological medical diagnoses
* Pregnant
* Severe medical diagnoses (e.g. cardiovascular, orthopedic)
* Skin allergies or irritation; open wounds
* Prisoners
* Cognitively impaired adults

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) amplitude during walking under each intervention condition | Day 1 (single study visit); Measured during each intervention condition (Assist, Resist, Sham)
  Muscle activation (specifically voltage amplitude) using wearable surface EMG of the gastrocnemius, lateral gastrocnemius, tibialis anterior, soleus, biceps femoris, rectus femoris, and gluteus maximus.

SECONDARY OUTCOMES:
6 Minute Walk Test | Day 1 (single study visit); Measured during each intervention condition (Assist, Resist, Sham)
  * The score of the test is the distance a patient walks in 6 minutes. Walking is self-paced on a standardized walk space using standardized instructions.
  * The patient may take as many standing rests as they like, but the timer should kept running and the number of rests taken and the total rest time recorded.
  * Assistive devices are allowed and must be documented.
  * Clinician assistance is permitted and must be from posterior so as not to pace the participant, and the level of assist must be documented.
  * When administering the test, do not walk in front of or directly beside the patient, as this may "pace" the patient and influence the speed and distance they walk. Instead, walk at least a half step behind the patient.
  * If a participant cannot walk but has goals and expectations to regain walking, a 6MWT score of 0 should be documented.
  * No talking should be done with the participant during the test other than the scripted and timed feedback outlined in the 6MWT guidelines.
10 Meter Walk Test | Day 1 (single study visit); Measured during each intervention condition (Assist, Resist, Sham)
  The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed). The distance covered is divided by the time it took the individual to walk that distance.
Gait Symmetry | Day 1 (single study visit); Measured during each intervention condition (Assist, Resist, Sham)
  Collect gait symmetry and other gait parameters such as stride length, using Kinect v2, GaitRite, and OpenCap. Kinect v2 tracks 3D joint kinematics to assess symmetry (left-right differences), stride length (foot displacement), and parameters like step time and velocity. GaitRite's pressure-sensitive walkway measures precise stride length, symmetry (step length/time differences), and parameters such as cadence and stance time. OpenCap, with multiple cameras and cloud processing, captures 3D kinematics to calculate symmetry, stride length, joint angles, and the Gait Deviation Index (GDI). Data will be synchronized, systems calibrated, and participants will walk naturally for analysis using dedicated software and scripts, ensuring comprehensive gait evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: James L Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab

IPD SHARING:
Plan to Share IPD: Yes